CLINICAL TRIAL: NCT03315780
Title: A Phase 4 Study to Evaluate Glucodynamic Effects of Dulaglutide in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of the Glucodynamic Effects of Dulaglutide (LY2189265) in Japanese Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 16730; H9X-JE-GBGK (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Results first posted 2019-04-30 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dulaglutide, Placebo (Experimental): Dulaglutide 0.75 mg administered subcutaneously (SC) once weekly for 4 weeks in period 1 followed by placebo administered SC once weekly for 4 weeks in Period 2. There is a 4 to 6 week washout period between Period 1 and Period 2.
  Interventions: Drug: Dulaglutide; Drug: Placebo
- Placebo, Dulaglutide (Experimental): Placebo administered SC once weekly for 4 weeks in Period 1 followed by Dulaglutide 0.75 mg administered SC for 4 weeks in Period 2. There is a 4 to 6 week washout period between Period 1 and Period 2.
  Interventions: Drug: Dulaglutide; Drug: Placebo

INTERVENTIONS:
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265
Drug: Placebo — Administered SC

SUMMARY:
The purpose of this study is to evaluate the glucodynamic effects of dulaglutide in Japanese participants with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes (based on the World Health Organization [WHO] diagnostic criteria) for at least 1 year.
* Have diet and exercise therapy only (no oral antihyperglycemic medication for at least 3 months prior to screening).
* Have a fasting blood glucose value of ≥120 and ≤200 milligrams per deciliter (mg/dL) at screening.
* Have a screening body weight of ≥50 and ≤80 kilograms.

Exclusion Criteria:

* Have known allergies to dulaglutide, or other glucagon-like peptide-1 (GLP-1) receptor agonists.
* Have had a clinically significant cardiovascular disease.
* Have a known clinically significant gastric emptying abnormality or have undergone gastric bypass surgery or restrictive bariatric surgery.
* Have acute or chronic hepatitis, signs and symptoms of any other liver disease.
* Have a history of chronic pancreatitis or acute idiopathic pancreatitis, or were diagnosed with any type of acute pancreatitis.
* Have an estimated glomerular filtration rate (eGFR) <30 milliliters/minute/1.73 meter squared.
* In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-28 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Inoue M, Shiramoto M, Oura T, Nasu R, Nakano M, Takeuchi M. Effect of Once-Weekly Dulaglutide on Glucose Levels in Japanese Patients with Type 2 Diabetes: Findings from a Phase 4, Randomized Controlled Trial. Diabetes Ther. 2019 Jun;10(3):1019-1027. doi: 10.1007/s13300-019-0605-7. Epub 2019 Apr 4. PMID 30949907

RESULTS

PARTICIPANT FLOW:
Groups:
- Dulaglutide Then Placebo: Dulaglutide 0.75 milligrams (mg) administered subcutaneously (SC) once weekly for 4 weeks in Period 1 followed by placebo administered SC once weekly for 4 weeks in period 2.
  There is a 4 to 6 week washout period between Period 1 and Period 2.
- Placebo Then Dulaglutide: Placebo administered SC once weekly for 4 weeks in Period 1 followed byDulaglutide 0.75 mg administered SC once weekly for 4 weeks in Period 2.
  There is a 4 to 6 week washout period between Period 1 and Period 2.
Period: Period 1
Arm/Group | Dulaglutide Then Placebo | Placebo Then Dulaglutide
Started | 6 | 6
Received One Dose of Study Drug | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Dulaglutide Then Placebo | Placebo Then Dulaglutide
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Overall: Participants were randomized to one of two treatment sequences: Dulaglutide 0.75 mg administered subcutaneously (SC) in Period 1 and placebo administered SC in Period 2 or placebo administered SC in Period 1 and Dulaglutide 0.75 mg administered in Period 2.
Arm/Group | Overall
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 12
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 12
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 8.5 (7.7)
Screening HbA1c [Mean (Standard Deviation); unit: percentage of HbA1c] | 7.9 (1.2)
Fasting Blood Glucose [Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)] | 164.67 (22.18)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glucose Area Under the Concentration Versus Time Curve From Time Zero to 4 Hours (AUC[0-4h])
Description: Least square (LS) means of glucose AUC 0-4h change from baseline was calculated using mixed-effects linear model. The model will include treatment, sequence, period, week, and treatment-by-week as fixed effects, baseline as a covariate, and participant as random effect.
Time Frame: Baseline, 4 Weeks
Population: All participants who receive at least one dose of study drug and have evaluable pharmacodynamic data.
Measure: Least Squares Mean (95% Confidence Interval); unit: milligram*hour per deciliter (mg*h/dL)
Groups:
- Dulaglutide: Dulaglutide 0.75 mg administered SC once weekly for four weeks.
- Placebo: Placebo administered SC once weekly for four weeks.
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 12
milligram*hour per deciliter (mg*h/dL) | -238.46 [-293.87 to -183.05] | 15.56 [-71.27 to 102.39]
Statistical Analysis 1: Comparison: Dulaglutide vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -254.02, 95% CI 2-sided [-337.76 to -170.28]

2. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Description: Change from baseline in fasting blood glucose obtained at pre-meal.
Time Frame: Baseline, 4 Weeks
Population: All participants who received at least one dose of study drug and evaluable had fasting blood glucose data.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 12
milligrams per deciliter (mg/dL) | -39.8 (33.3) | -8.2 (21.5)

3. Secondary Outcome: Change From Baseline in Postprandial Blood Glucose
Description: Change from baseline in postprandial blood glucose at 120 minutes at week 4.
Time Frame: Baseline, 4 Weeks
Population: All participants who received at least one dose of study drug and had evaluable postprandial blood glucose data.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 12
mg/dL | -67.0 (32.1) | 13.9 (28.7)

4. Secondary Outcome: Change From Baseline in Insulin Area Under the Concentration Versus Time Curve From Time Zero to 4 Hours (AUC [0-4h])
Description: LS mean of the insulin change from baseline was analyzed using a mixed-effects linear model. The model includes treatment, sequence, period, week and treat-by-sequence as fixed effects, baseline as a covariate and participant as random effect.
Time Frame: Baseline, 4 Weeks
Population: All participants who received at least one dose of study drug and had evaluable insulin data.
Measure: Least Squares Mean (95% Confidence Interval); unit: insulin units*h/mL (µU*h/mL)
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 12
insulin units*h/mL (µU*h/mL) | 25.20 [7.29 to 43.10] | -2.27 [-11.39 to 6.85]
Statistical Analysis 1: Comparison: Dulaglutide vs Placebo; Test type: Superiority; p = 0.0100, Mixed Models Analysis; Mean Difference (Final Values) = 27.46, 95% CI 2-sided [8.05 to 46.87]

5. Secondary Outcome: Change From Baseline in C-Peptide Area Under the Concentration Versus Time Curve From Time Zero to 4 Hours (AUC [0-4h])
Description: LS mean of C-peptide change from baseline was analyzed using a mixed-effects linear model. The model includes treatment, sequence, period, week and treat-by-sequence as fixed effects, baseline as a covariate and participant as random effect.
Time Frame: Baseline, 4 Weeks
Population: All participants who received at least one dose of study drug and had evaluable c-peptide data.
Measure: Least Squares Mean (95% Confidence Interval); unit: nanogram*h/milliliter (ng*h/mL)
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 12
nanogram*h/milliliter (ng*h/mL) | 3.58 [0.44 to 6.72] | -0.14 [-1.24 to 0.96]
Statistical Analysis 1: Comparison: Dulaglutide vs Placebo; Test type: Superiority; p = 0.0263, Mixed Models Analysis; Mean Difference (Final Values) = 3.72, 95% CI 2-sided [0.63 to 6.81]

6. Secondary Outcome: Change From Baseline in Glucagon Area Under the Concentration Versus Time Curve From Time Zero to 4 Hours (AUC [0-4h])
Description: LS mean of glucagon change from baseline was analyzed using a mixed-effects linear model. The model includes treatment, sequence, period, week and treat-by-sequence as fixed effects, baseline as a covariate and participant as random effect.
Time Frame: Baseline, 4 Weeks
Population: All participants who received at least one dose of study drug and had evaluable glucagon data.
Measure: Least Squares Mean (95% Confidence Interval); unit: picomole*h/Liter (pmol*h/L)
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 12
picomole*h/Liter (pmol*h/L) | -16.39 [-25.69 to -7.09] | -7.02 [-12.81 to -1.24]
Statistical Analysis 1: Comparison: Dulaglutide vs Placebo; Test type: Superiority; p = 0.0800, Mixed Models Analysis; Mean Difference (Final Values) = -9.36, 95% CI 2-sided [-20.16 to 1.43]

7. Secondary Outcome: Change From Baseline in Triglyceride Area Under the Concentration Versus Time Curve From Time Zero to 4 Hours (AUC [0-4h])
Description: LS mean of triglyceride change from baseline was analyzed using a mixed-effects linear model. The model includes treatment, sequence, period, week and treat-by-sequence as fixed effects, baseline as a covariate and participant as random effect.
Time Frame: Baseline, 4 Weeks
Population: All participants who received at least one dose of study drug and had evaluable triglyceride data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg*h/dL
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 12
mg*h/dL | 31.02 [-54.70 to 116.74] | 46.41 [-76.55 to 169.38]
Statistical Analysis 1: Comparison: Dulaglutide vs Placebo; Test type: Superiority; p = 0.7475, Mixed Models Analysis; Mean Difference (Final Values) = -15.39, 95% CI 2-sided [-118.35 to 87.57]

8. Secondary Outcome: Number of Participants Who Develop Hypoglycemic Events
Description: Number of participants who develop hypoglycemic events.
Time Frame: Baseline through 4 weeks
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 14 weeks
Description: All participants who received at least one dose of study drug.
Arm/Group | Dulaglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dulaglutide (N=12) | Placebo (N=12)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Pericoronitis (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT03315780/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT03315780/SAP_001.pdf